CLINICAL TRIAL: NCT03256422
Title: Randomized, Open-label and Multicentric Trial Evaluating the Non-inferiority of Antiretroviral Treatment Taken 4 Consecutive Days Per Week Versus Continuous Therapy 7/7 Days Per Week in HIV-1 Infected Patients With Controlled Viral Load Under Antiretroviral Therapy
Brief Title: Antiretroviral Treatment Taken 4 Days Per Week Versus Continuous Therapy 7/7 Days Per Week in HIV-1 Infected Patients
Acronym: QUATUOR
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: IMEA Leon M'Ba Foundation (Unknown); INSERM UMR S 1136 (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANRS 170 - QUATUOR
Record Dates: First submitted 2017-08-09; First posted 2017-08-22 (Actual); Last update posted 2018-02-05 (Actual); Status verified 2017-08

CONDITIONS: HIV Infections
Keywords: Controlled, virological and therapeutic success, treatment discontinution, 4 days per week
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Intervention Model Description: Open-label, randomized trial in 2 parallel groups
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 4 days / 7 (Experimental): Patients included in this arm will take their ARV treatment 4 consecutive days per week during 98 weeks
  Interventions: Drug: Treatment discontinuation
- 7 days / 7 (Active Comparator): Patients included in this arm will continue their ARV therapy 7 days per weeks during 48 weeks and after W48, they will take their ARV treatment 4 days per week until W98
  Interventions: Drug: Treatment discontinuation

INTERVENTIONS:
Drug: Treatment discontinuation — • Receiving tritherapy. Allowed treatment drugs are :
  1. nucleoside analogs : tenofovir (TDF ou TAF), emtricitabine, abacavir, lamivudine
  2. protease inhibitors : lopinavir/r, darunavir/r ou atazanavir/r
  3. non nucleoside reverse transcriptase inhibitors : efavirenz, rilpivirine ou etravirine
  4. integrase inhibitors : dolutegravir, elvitegravir/cobicistat ou raltegravir

SUMMARY:
The trial is an open-label, multicenter, prospective, randomized trial in 2 parallel groups, evaluating at W48, the non-inferiority of antiretroviral treatment taken 4 consecutive days a week versus continuous therapy, in HIV infected patients with controlled viral load for at least 12 months and stable antiretroviral treatment since 4 months.

DETAILED DESCRIPTION:
Open-label, multicenter, prospective, randomized trial in 2 parallel groups, evaluating at W48, the non-inferiority of antiretroviral treatment taken 4 consecutive days a week versus continuous therapy, in HIV infected patients with controlled viral load for at least 12 months and stable antiretroviral treatment since 4 months. The non-inferiority margin (delta) is 5%. The randomization will be stratified according to the family of the third antiretroviral agent (II, PI, and NNRTI). A minimum of 200 patients will be included in the integrase inhibitor strata to provide a sufficient power to assess the efficacy of strategy in this population.

At W48, all patients with virological success in the continuous therapy group will switch to the 4/7 days therapy.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection, coinfection HIV-1/HIV-2 possible
* Age≥18 years old
* Current therapy unchanged for the last 4 months
* Receiving tritherapy with 2 nucleoside reverse transcriptase inhibitor+protease inhibitors or 2 nucleoside reverse transcriptase inhibitor+non-nucleoside reverse transcriptase inhibitors or 2 nucleoside reverse transcriptase inhibitor+integrase inhibitors.

Allowed treatment drugs are :

1. nucleoside analogs : tenofovir (TDF ou TAF), emtricitabine, abacavir, lamivudine 2. protease inhibitors : lopinavir/r, darunavir/r ou atazanavir/r 3. Non nucleoside reverse transcriptase inhibitors : efavirenz, rilpivirine ou etravirine 4. integrase inhibitors : dolutegravir, elvitegravir/cobicistat ou raltegravir

* Viruses susceptible to all antiretroviral drugs present in the ongoing tritherapy (AC11-ANRS algorithm).

  1. If a genotype is available in the patient medical history; viruses must be susceptible to all ongoing antiretroviral drugs
  2. If no RNA genotype available, a genotype will be performed on DNA at screening and will not have to show any resistance to the ongoing antiretroviral drugs
* Viral load (VL) < 50 cp/mL in the past year, with at least 3 VL measurements including screening; only one episode of viral blip < 200 copies/mL is authorized in the last year
* CD4 T cells > 250/mm3 at the screening visit
* Estimated glomerular filtration rate > 60 mL/min (Chronic Kidney Disease - Epidemiology Collaboration method)
* Transaminases : aspartate aminotransférase et alanine aminotransférase < 3N
* Haemoglobin > 10 g/dL
* Platelets > 100 000/mm3
* For women of childbearing age, negative pregnancy test at screening; agree to use mechanical contraception during the study
* Social security system coverage
* Informed consent form signed by patient and investigator

Exclusion Criteria:

* Infection by HIV-2
* Chronic and active Viral B Hepatitis with positive antigen HBs
* Chronic and active Viral C Hepatitis with treatment expected in the next 98 weeks
* Concomitant treatment using interferon, interleukins, any other immune-therapy or chemotherapy, antivitaminK for patients on ARVT using a booster
* Concomitant prophylactic or curative treatment for an opportunistic infection
* All conditions (use of alcohol, drugs, etc.) judged by the investigator to possibly interfere with study protocol compliance, observance and/or study treatment tolerance
* Pregnant or breast feeding women
* Subjects under "sauvegarde de justice" (judicial protection due to temporarily and slightly diminished mental or physical faculties), or under legal guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 640 (Estimated)
Dates: Start 2017-09-07 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with therapeutic success at Week 48. | Week 48
  To evaluate after 48 weeks the therapeutic success of a weekly strategy of 4 consecutive days on treatment followed by 3 days off treatment, defined by :
  * absence of virological failure : a measure of the viral load will be done, this measure have to be < 50 cp/mL. If it's > 50 cp/mL, a second measure will be done at 2 to 4 weeks apart. If it's still > 50 cp/mL, it's a virological failure
  * no discontinuation or modification of the study strategy for more than 30 consecutive days.

SECONDARY OUTCOMES:
Proportion of patients with therapeutic success at Week 96 | Week 96
  To evaluate after 96 weeks the therapeutic success of a weekly strategy of 4 consecutive days on treatment followed by 3 days off treatment, defined by :
  * absence of virological failure : a measure of the viral load will be done, this measure have to be < 50 cp/mL. If it's > 50 cp/mL, a second measure will be done at 2 to 4 weeks apart. If it's still > 50 cp/mL, it's a virological failure
  * no discontinuation or modification of the study strategy for more than 30 consecutive days.
Virological success | Week 48 and Week 96
  The HIV-1 viral load at week 48 must be inferior to 50 copies/mL
Number of virological " blips " | between Week 0 and Week 48, and between Week 0 and Week 96
  viral load > 50 copies/mL followed by a control value ≤ 50 cp/mL
Percentage of patients with a viral load signal detected | between Week 0 and Week 48 and Week 0 and Week 96
  (subgroup of patients tested with Roche-Taqman, threshold<20 copies/mL)
Proportion of patients with acquisition of drugs resistance mutations in case of virological failure detected by Sanger and by next generation sequencing | Week 4, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 96 (if it's necessary)
Frequency of minority resistant variants archived in DNA at Week 0 and their impact on virological failure (2 consecutive VL> 50 copies / mL) and on the acquisition of drugs resistance mutations | Week 0
Evolution of ultra sensitive viral load and total DNA in the peripheral blood mononuclear cells at Week 0, Week 24, Week 48 and Week 96; evolution of viral genotypic sequence between Week 0, Week 48 and Week 96 (subgroup of 120 patients) | between Week 0, Week 48 and Week 96
  Immuno-viro-pharmacological sub-study of 120 patients
Description of the factors associated with virological rebound (viral load >50 cp/mL). | Week 4, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 96 (if it's necessary)
  (viral load >50 cp/mL).
Evolution of T cluster of differentiation 4 and cluster of differentiation 8 cells count, and T cluster of differentiation 4 /cluster of differentiation 8 ratio | from Week-4 to Week 48 and Week 96
  Measurement of T cluster of differentiation 4 cell count, T cluster of differentiation 8 cell count, and T cluster of differentiation 4 /T cluster of differentiation 8 ratio
Evolution of fasting metabolic parameters | until Week 48 and Week 96
  Measurement of total cholesterol total, LDL-C, HDL-C, Triglycerides and glycemia
Evolution of inflammation and immune activation parameters | from Week 0 to Week 24 and Week 48
  Measurement of sCD14, sCD163, IP-10, C-reactive protein, interleukin-6 et D-dimerus, soluble TNF receptor 1, soluble TNF receptor 2 Immuno-viro-Pharmacological Sub-study in 120 patients
HIV RNA viral load in semen | Week 0, Week 24 and Week 48
  Sperm sub-study (120 patients)
Residual plasmatic concentrations of the third antiretroviral agent | Week 0, Week 4, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84 and Week 96
  Measurement of the third antiretroviral agent plasmatic concentration (protease inhibitors or non-nucleoside reverse transcriptase inhibitors or integrase inhibitors)
Residual plasmatic concentrations of tenofovir (TDF or TAF) | Week 0, Week 4, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84 and Week 96
  Measurement of tenofovir plasmatic concentration
Residual intracellular concentrations of the third antiretroviral agents | Week 0, Week 24 and Week 48
  Immuno-viro-Pharmacological sub-study (120 patients) Measurement of the third antiretroviral agent intracellular concentration (protease inhibitors or non-nucleoside reverse transcriptase inhibitors or integrase inhibitors)
Treatment adherence | Week 0, Week 12, Week 24, Week 36, Week 48, Week 72,and Week 96
  Evaluation by a self-reported questionnaire
Quality of life | Week-4, Week 0, Week 48 and Week 96
  Evaluation by a self-reported questionnaire
Patient satisfaction | Week 0, Week 12, Week 48 and Week 96
  Evaluation by a self-reported questionnaire
Pharmaco-economic aspects of the strategy | Between Week 0 and Week 98
  Assessment and comparison of cost essay between each arm.
Median time to virologic failure | Between week 0 and 98
  Measure the delay between week 0 and the date of different virologic failure
Frequency of grade 3 or more adverse events, adverse effects, drug-modifying adverse events, drug-related adverse events and serious adverse events (SAE) | Between Week 0 and Week 98
  according to the sponsor's grading scale

CONTACTS AND LOCATIONS:
Overall Officials: Pierre De Truchis, MD, Principal Investigator — Hôpital Raymond Poincaré
Locations (63):
- France (63):
  - CHU Pointe-à-Pitre, Pointe à Pitre, Guadeloupe
  - Hôpital La Meynard Zobda Quitman, Fort-de-France, Martinique
  - Centre hospitalier Victor Dupouy, Argenteuil
  - Hôpital Henri Duffaut, Avignon
  - CHRU Jean Minjoz, Besançon
  - Avicenne, Bobigny
  - Jean Verdier, Bondy
  - Hôpital Saint-André, Bordeaux
  - Hôpital Pellegrin, Bordeaux
  - Hôpital Ambroise Paré, Boulogne-Billancourt
  - Hôpital de la Côte de Nacre, Caen
  - Hôpital Louis Pasteur, Chartres
  - Antoine Beclère, Clamart
  - Hôpital Gabriel Montpied, Clermont-Ferrand
  - Centre hospitalier sud francilien, Corbeil-Essonnes
  - CHI de Créteil, Créteil
  - Hôpital Henri Mondor, Créteil
  - Hôpital du Bocage, Dijon
  - Hôpital Raymond Poincaré, Garches
  - Hôpital Michallon, Grenoble
  - CHD de la Roche Sur Yon, La Roche-sur-Yon
  - Bicêtre, Le Kremlin-Bicêtre
  - Centre Hospitalier du Mans, Le Mans
  - Institut hospitalier franco-britannique, Levallois-Perret
  - Hôpital Dupuytren, Limoges
  - Hôpital de la Croix Rousse, Lyon
  - Hôpital Edouard Herriot, Lyon
  - Hôpital Sainte Marguerite, Marseille
  - Hôpital Européen, Marseille
  - Hôpital Gui de Chauliac, Montpellier
  - Hôpital Emile Müller, Mulhouse
  - Hôpital de l'Hôtel Dieu, Nantes
  - Hôpital de l'Archet, Nice
  - Hôpital Carémeau, Nîmes
  - Hôpital de La Source, Orléans
  - Hôpital Saint-Antoine, Paris
  - Hôpital Necker, Paris
  - Hôpital Bichat, Paris
  - Hôpital de l'Hôtel Dieu, Paris
  - Hôtel-Dieu, Paris
  - Hôpital Saint-Louis, Paris
  - Lariboisière, Paris
  - Hôpital Pitié-Salpêtrière, Paris
  - Hôpital Européen Georges Pompidou, Paris
  - Tenon, Paris
  - Centre Hospitalier de Perpignan, Perpignan
  - Centre Hospitalier René Dubos, Pontoise
  - Centre hospitalier Annecy Genevois, Pringy
  - Hôpital Robert Debré, Reims
  - Hôpital Pontchaillou, Rennes
  - Centre Hospitalier de Saint-Brieuc, Saint-Brieuc
  - Hôpital Delafontaine, Saint-Denis
  - Hôpital Nord, Saint-Etienne
  - Centre Hospitalier Général de Saint Nazaire, Saint-Nazaire
  - Hôpital Civil, Strasbourg
  - Hôpital Foch, Suresnes
  - Hôpital La Grave, Toulouse
  - Hôpital Purpan, Toulouse
  - Hôpital Gustave Dron, Tourcoing
  - Hôpital Bretonneau, Tours
  - Hôpital de Brabois, Vandœuvre-lès-Nancy
  - Hôpital André Mignot, Versailles
  - Centre Hospitalier Intercommunal, Villeneuve-Saint-Georges

REFERENCES:
- [Derived] Landman R, de Truchis P, Assoumou L, Lambert S, Bellet J, Amat K, Lefebvre B, Allavena C, Katlama C, Yazdanpanah Y, Molina JM, Petrov-Sanchez V, Gibowski S, Alvarez JC, Leibowitch J, Capeau J, Fellahi S, Duracinsky M, Morand-Joubert L, Costagliola D, Alvarez JC, Girard PM; ANRS 170 QUATUOR study group. A 4-days-on and 3-days-off maintenance treatment strategy for adults with HIV-1 (ANRS 170 QUATUOR): a randomised, open-label, multicentre, parallel, non-inferiority trial. Lancet HIV. 2022 Feb;9(2):e79-e90. doi: 10.1016/S2352-3018(21)00300-3. PMID 35120640